CLINICAL TRIAL: NCT00389701
Title: Phase II Trial of Twice Weekly Induction Followed by Once Weekly IV Velcade (Bortezomib) With Dexamethasone in Patients With Relapsed and/or Refractory Multiple Myeloma Following at Least 1 Prior Therapy
Brief Title: Bortezomib and Dexamethasone in Treating Patients With Multiple Myeloma That Has Relapsed or Has Not Responded to Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sparrow Regional Cancer Center (Other)
Responsible Party: Gordan Srkalovic, Sparrow Regional Cancer Center
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000509044; SPARROW-I071-341-03; SPARROW-IRB-6016
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Dexamethasone

INTERVENTIONS:
Drug: bortezomib
Drug: dexamethasone

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with dexamethasone may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with dexamethasone works in treating patients with multiple myeloma that has relapsed or has not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall response rate (complete response and partial response) in patients with relapsed or refractory multiple myeloma treated with induction therapy and maintenance therapy comprising bortezomib and dexamethasone.

Secondary

* Determine the toxicity of this regimen in these patients
* Determine the tolerability of this regimen in these patients.
* Determine the duration of response in patients treated with this regimen.
* Determine time to progression in patients treated with this regimen.
* Determine overall and progression-free survival of patients treated with this regimen.

OUTLINE: This is an open-label study.

* Induction therapy: Patients receive bortezomib IV on days 1, 4, 8, and 11. Patients also receive oral dexamethasone on days 1, 2, 4, 5, 8, 9, 11, and 12. Treatment repeats every 21 days for 4 courses. Patients who achieve complete response (CR) receive an additional 2 courses of induction therapy and proceed to maintenance therapy.
* Maintenance therapy: Patients receive bortezomib IV on days 1, 8, 15, and 22. Patients also receive oral dexamethasone on days 1, 2, 8, 9, 15, 16, 22, and 23. Treatment repeats every 36 days in the absence of disease progression or unacceptable toxicity. Patients who achieve CR receive an additional 2 courses of maintenance therapy beyond documentation of CR.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  * Refractory or relapsed disease meeting the following criteria:

    * Primary refractory disease and first-line relapsing disease
    * Progressive disease after last therapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Platelet count ≥ 50,000/mm³ (≥ 30,000/mm³ for patients with significant bone marrow involvement)

  * Transfusions allowed
* Hemoglobin ≥ 7.5 g/dL
* Absolute neutrophil count ≥ 750/mm³
* Serum calcium < 14 mg/dL
* AST and ALT < 2.5 times upper limit of normal
* Creatinine clearance ≥ 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No peripheral neuropathy ≥ grade 2 within the past 14 days
* No hypersensitivity to boron or mannitol
* No cardiovascular complications, including any of the following:

  * Myocardial infarction within the past 6 months
  * New York Heart Association class III-IV heart failure
  * Uncontrolled angina
  * Ventricular arrhythmias
  * Electrocardiographic evidence of acute ischemia or active conduction system abnormalities
  * Cardiac amyloidosis
* No other cancer or treatment for cancer other than basal cell cancer of the skin within the past 5 years
* No poorly controlled chronic diseases (e.g., diabetes mellitus or hypertension)
* No HIV positivity
* No hepatitis B surface antigen or active hepatitis C infection
* No active systemic infection requiring therapy
* No serious medical or psychiatric illness that would interfere with study participation

PRIOR CONCURRENT THERAPY:

* No plasmapheresis within the past 4 weeks
* No major surgery within the past 4 weeks
* No prior bortezomib
* No chemotherapy (e.g., clarithromycin) within the past 4 weeks
* No radiotherapy within the past 3 weeks
* No corticosteroids (> 10 mg/day of prednisone or equivalent) within the past 3 weeks
* No other immunotherapy within the past 8 weeks
* No other investigational drugs within the past 14 days
* No concurrent participation in other clinical research studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Toxicity
Tolerability
Duration of response after completion of treatment
Time to progression
Overall and progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Gordan Srkalovic, MD, PhD, Study Chair — Sparrow Regional Cancer Center
Locations (1):
- Sparrow Regional Cancer Center, Lansing, Michigan, United States